CLINICAL TRIAL: NCT05801588
Title: T'ai Chi Mild Exercise: The Potential for Reducing Pain and Improving Quality of Life Among Those With Back Pain
Brief Title: Participating in T'ai Chi to Reduce Back Pain and Improve Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMB15574
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Low Back Pain
Keywords: T'ai Chi; Qigong
MeSH Terms: conditions — Low Back Pain | interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T'ai Chi and Qigong Rehabilitation (Experimental): T'ai chi/Qigong is a multidimensional (mind, body, and spirit integrative) and multimodal (strength, flexibility, balance, posture, and light to moderate aerobic) form of exercise that is safe for persons of all ages and physical abilities. The 12-week, twice-per-week t'ai chi and qigong gentle movement and meditation program proposed to be studied is adapted from the WaQi program, a curriculum developed by Master Yang Yang, PhD. The practice is gentle yet powerful, aiming to relieve and prevent back, neck, and hip pain. It has an online teaching module and is uniquely suited for our study population. The program requires no difficult movement transitions, but still contains all essential parts including meditation. The WaQi program has less psychological stress and physical challenge than other exercise activities because it can be performed either sitting, standing, and lying down.
  Interventions: Other: T'ai Chi and Qigong Rehabilitation
- Usual care (Active Comparator): The control arm will receive the same 12-week, twice-per-week t'ai chi and qigong gentle movement and meditation, online live T'ai Chi and Qigong teaching module from Jan. 26, 2023 to April 17, 2023.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: T'ai Chi and Qigong Rehabilitation — T'ai chi/Qigong is a multidimensional (mind, body, and spirit integrative) and multimodal (strength, flexibility, balance, posture, and light to moderate aerobic) form of exercise that is safe for persons of all ages and physical abilities. The 12-week, twice-per-week t'ai chi and qigong gentle movement and meditation program proposed to be studied is adapted from the WaQi program, a curriculum developed by Master Yang Yang, PhD. The practice is gentle yet powerful, aiming to relieve and prevent back, neck, and hip pain. It has an online teaching module and is uniquely suited for our study population. The program requires no difficult movement transitions, but still contains all essential parts including meditation. The WaQi program has less psychological stress and physical challenge than other exercise activities because it can be performed either sitting, standing, and lying down.
  Arms: T'ai Chi and Qigong Rehabilitation
Other: Usual care — The control arm will receive the same 12-week, twice-per-week t'ai chi and qigong gentle movement and meditation, online live T'ai Chi and Qigong teaching module from Jan. 26, 2023 to April 17, 2023.
  Arms: Usual care

SUMMARY:
The purpose of the study is to examine the implementation strategy, in terms of feasibility and the possible benefits, of a free online Zoom t'ai chi and qigong gentle movement and meditation program to reduce back pain and improve sleep and quality of life among those with chronic back pain. The primary objective of this study is to examine whether a safe and moderate online t'ai chi and qigong exercise program, offered without cost to individuals with chronic back pain, improves pain levels, sleep, and quality of life; The secondary objective is to explore whether improvements in pain levels are different among smokers and those with unhealthy BMI than among others.

DETAILED DESCRIPTION:
The purpose of the study is to examine the implementation strategy, in terms of feasibility and the possible benefits, of a free online Zoom t'ai chi and qigong gentle movement and meditation program to reduce back pain and improve sleep and quality of life among those with chronic back pain. The primary objective of this study is to examine whether a safe and moderate online t'ai chi and qigong exercise program, offered without cost to individuals with chronic back pain, improves pain levels, sleep, and quality of life; The secondary objective is to explore whether improvements in pain levels are different among smokers and those with unhealthy BMI than among others.

Study Design and Methods:

The study will be a prospective, randomized controlled trial with two groups: a t'ai chi and qigong exercise (treatment) group and a waitlist control group. The waitlist control group will simply be a comparison group.

The study team will conduct a single-centered, single-blind, parallel design, randomized controlled trial with 300 participants randomly allocated to one of two arms: a waitlist control or a 12-week, twice per week, T'ai Chi and Qigong exercise.

Consent for participation in the t'ai chi gentle movement and meditation program and completion of the baseline and three additional surveys will be included in the Survey. The Informed Consent for participation in the study will be prompted before the start of the initial Survey in Qualtrics. Potential participants of the t'ai chi classes cannot advance to the survey or participate in the t'ai chi program without accepting consent for participation. In the event consent is declined, the survey is prompted to end.

Statistical methods: The study will be a prospective, randomized controlled trial with two groups: a t'ai chi and qigong exercise (treatment) group and a waitlist control group. The treatment group started the t'ai chi and qigong classes in September 2022; the waitlist group was offered instruction beginning in January 2023. The waitlist control group will simply be a comparison group. Thus, we will be comparing the outcomes of key measures between the treatment group receiving t'ai chi and qigong instruction starting in September and the waitlist control group.

After the baseline survey was closed to further responses, the data was exported as an SPSS file, then converted to Stata, by the PI onto his NYMC-issued, password-protected computer, which is in a secure space. Participants then were randomized either to start class in September 2022 (the treatment group) or January 2023 (the waitlisted control group).

The treatment and waitlist control groups were randomized using Stata statistical software through a standard randomization algorithm. The algorithm would ensure that participants had an equal chance of being assigned to either arm. A simple, post-randomization analysis of participants assigned to the two arms was conducted to confirm that participants in the treatment and control groups are similar in terms of baseline Oswestry Disability Index (ODI) scores. (A comparison of means t-test will be used.)

Previously validated, self-administered survey instruments will be included in the Survey to be used to assess the primary outcome of interest, low back pain, as well as associated outcomes of sleep and quality of life, including:

* The Oswestry Disability Index (primary pain measurement)
* The Visual Analog Scale for Back and Leg Pain (additional pain measurement)
* The "SF-36," Short Form Health Survey questionnaire (health and quality of life)
* 19-Item Pittsburgh Sleep Quality Index

A maximum of 300 people with chronic low back pain were selected to participate in the program on a first-come basis. The treatment and control groups were divided into roughly equal numbers, with a maximum of 150 participants selected for participation in the live Zoom t'ai chi classes starting in September 2022 and a maximum of 150 participants selected for the waitlist control. The project will include a minimum of 200 total recruited participants, which, accounting for possible attrition, will result in a minimum of 50 participants in each study group, enough to statistically analyze the primary outcome of pain alleviation (see Sample Size and Power below).

Statistical comparisons of the treatment and waitlist control group will be based on four surveys:

* Baseline survey sent three weeks before the start of September 2022 of the t'ai chi and qigong gentle movement and mediation class. The survey closed one week prior to class start.
* Intermediate survey sent after Week 8 of the September start.
* Post-intervention survey sent the day after the last of the classes that started in September (that is, after the 24th class).
* Follow-up survey sent four weeks later.

Separate statistical tests will be run by secondary variables of interest, including smoking status and BMI; specifically, the main outcomes of interest (pain, sleep, and quality of life) will be cross-tabulated by the secondary variables. Similar statistical comparisons will be made between pain levels and sleep, and between pain levels and quality of life measures. A Fisher's exact test will be applied to test the statistical significance of such cross-tabulated variables.

Descriptive statistics of all pertinent measures of all participants, as well as simple correlation matrices, will also be included in our analysis.

At the completion of the intervention/study, 25 qualitative interviews will be conducted to assess the barriers and facilitators related to implementing the online T'ai Chi and Qigong intervention.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years and over
* Have experienced low back pain for the last 6 weeks or longer
* Understands written and spoken English
* Be willing to complete the initial survey and 3 additional ones emailed baseline and January 2023
* Be willing and able to provide consent to participate in the survey

Exclusion Criteria:

* Excluded if pregnant
* Excluded if subject previously has taken t'ai chi classes
* Excluded if subject has had spine surgery within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
Change in ODI 3 months after intervention | baseline, 3 months
  The Oswestry Disability Index (ODI) is a commonly used outcome measure for individuals with low back pain. The ODI includes 10 questions about pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and traveling, each based upon a 6-item Likert scale. Each section is scored on a 0-5 scale, 5 representing the greatest disability. If a respondent does not answer all 10 questions, then average scores and levels of disability are adjusted to account for skipping. If all 10 questions are answered, then the maximum score possible is 50 (10 x 5); if 9 are answered, then the maximum score is 45 (9 x 5), and so on. Someone with a total score of 18 out of a maximum of 50 (all 10 questions answered) would have a percentage score of 18/50 = 35%. A score of 18 out of 45 (9 questions answered) would result in a percentage score of 18/45 = 40%. Categories of disability range from minimal, moderate, severe, crippled, and bed-bound.

SECONDARY OUTCOMES:
Change in VAS back pain | baseline, 3 months
  The visual analog scale (VAS) is a validated, subjective measure of pain that is commonly used in research. The VAS measures pain intensity on a scale of 0 to 10, with 0 representing no pain and 10 representing the worst pain imaginable.
Change in VAS leg pain | baseline, 3 months
  The visual analog scale (VAS) is a validated, subjective measure of pain that is commonly used in research. The VAS measures pain intensity on a scale of 0 to 10, with 0 representing no pain and 10 representing the worst pain imaginable.
The "SF-36," Short Form Health Survey questionnaire | baseline, 3 months
  The "SF-36," Short Form Health Survey questionnaire (health and quality of life) a widely used tool for assessing Health-Related Quality of Life. The SF-36 assesses eight scales: (1) Physical functioning, (2) Role limitations due to physical health, (3) Role limitations due to emotional problems, (4) Energy/fatigue, (5) Emotional well-being, (6) Social functioning, (7) Pain, and (8) General health. For each of these eight scales, the lower the score, the greater the indication of disability. A score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. The following ranges are used as guideline values for categorizing the level of disability: Severe disability = 0-24.99; Moderate disability = 25-49.99; Mild disability = 50-74.99; and Minimal to no disability = 75-100.
19-Item Pittsburgh Sleep Quality Index | baseline, 3 months
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score (range 0-21), where a higher score corresponds to lower sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A Knapp, PhD, Principal Investigator — New York Medical College, Valhalla, NY 10595
Locations (1):
- New York Medical College, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: Data requests can be submitted starting 12 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following the review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact kenneth_knapp@nymc.edu

REFERENCES:
- [Derived] Yang Y, McCluskey S, Bydon M, Singh JR, Sheeler RD, Nathani KR, Krieger AC, Mehta ND, Weaver J, Jia L, DeCelle S, Schlagal RC, Ayar J, Abduljawad S, Stovitz SD, Ganesh R, Verkuilen J, Knapp KA, Yang L, Hartl R. A Tai chi and qigong mind-body program for low back pain: A virtually delivered randomized control trial. N Am Spine Soc J. 2024 Sep 8;20:100557. doi: 10.1016/j.xnsj.2024.100557. eCollection 2024 Dec. PMID 39469294